CLINICAL TRIAL: NCT04571905
Title: "Magnesium-based, Bioresorbable Implants for Pediatric Elbow Fractures, a Single Center Pilot Study for Osteosynthesis With Magnezix Screws in Fractures of the Epicondylus Ulnaris and Condylus Radialis."
Brief Title: MagnezixKids Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Krebs (Other)
Responsible Party: Sponsor-Investigator, Thomas Krebs, Surgeon in Chief, Member of the executive board, Ostschweizer Kinderspital
Organization: Ostschweizer Kinderspital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTU 18.028
Record Dates: First submitted 2020-08-11; First posted 2020-10-01 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Magnesium-based; Bioresrobable Implants; Pediatric Elbow Fractures; Osteosynthesis; Childhood; Magnezix; Elbow Fracture
MeSH Terms: conditions — Elbow Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Syntellix Treatment Arm (Other): General anaesthesia, open fracture reduction, insertion of the appropriate screw with x-ray control and documentation intraoperatively, cast immobilisation Use of bioresorbable Magnezix CS or CBS Screws, if intraoperatively suitable bioresorbable screws not available, use of conventional ostesynthesis screws
  Interventions: Device: Osteosynthesis with resorbable Material

INTERVENTIONS:
Device: Osteosynthesis with resorbable Material — Osteosynthesis with Magnezix screws in fractures of the Epicondylus ulnaris and Condylus radialis under General anaesthesia
  Other Names: Magnezix (Syntellix) screws

SUMMARY:
The overall objective of the study is to describe the outcomes of osteosyn-thesis with magnesium based screws in children with a primary or second-ary (within 7 days from trauma) dislocated fracture of the Epicondyles ul-naris or Condylus radialis, and to compare them with outcomes of conven-tional osteosynthesis using steel screws.

If our results suggest non-inferiority of osteosynthesis with magnesium-based screws, the procedure could be tested formally in a subsequent full-size study.

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary (within 7 days from trauma) dislocated fracture of the Epicondyles ulnaris or Condylus radialis (indication for operative treatment according to international standard: Dislocation of more than 2 mm in Condylus radials fractures and more than 5 mm in Epicondylus ulnas fractures )
* Age 3-15 years
* Informed Consent as documented by signature

Exclusion Criteria:

* - open fractures or complex multi fragment fractures that require dif-ferent osteosynthetic procedures than screw fixation
* severe local accompanying injury (injury to nerves/vessels)
* polytrauma patients
* fracture age > 7 days
* preexisting ipsilateral elbow fracture
* relevant comorbidities, which have influence on fracture and wound healing
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant or the legal representatives
* Previous enrolment into the current study
* Enrolment of the investigator's family members and other dependent persons
* Any of the following applicable absolute and relative contraindica-tions listed in the MAGNEZIX® CBS and CSc 4.8 mm instruction for use :

Absolute contraindications:

* insufficient or avascular bone mass for anchorage of the implant, ex-cept osteochondral fractures and dissecates
* confirmation or suspected septic infectious surgical site
* application in the area of the epiphyseal plates

Relative contraindications:

* acute sepsis
* alcohol, nicotine and/or drug abuse
* epilepsy
* poor skin/soft tissue conditions
* uncooperative patient or patient with restricted intellectual capacity
* no options for adequate postoperative treatment (e.g. temporary strain relief)

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Clinical and radiologic outcome (fracture consolidation) | 12 months
  radiologic outcome after osteosynthesis with magnesium based screws in children with a primary or secondary (within 7 days from trauma) dislocated fracture of the Epicondyles ulnaris or Condylus radialis Fracture alignment is measured as dislocation distance (mm). Appropriate alignement is a postopera-tive dehiscence or dislocation of less than 5 mm in Epicondylus ulnaris fractures and less than 2 mm in Condylus radialis fractures, according to literature (26/27/31).

SECONDARY OUTCOMES:
Analgesic reuirement | 12 months
  Analgesic requirement via Pain score (Visual Analog Scale, VAS, Range from 1 (no pain) to 10 (strongest pain)) (27) at every study visit (except visit 1: preop. assessment)
ROM | 12 months
  Clinical reassessment at Routine follow-ups at every study visit
  - An Arc >100° shows a good functional result, arc 50-100° is a fair (acceptable) result, arc <50° shows a poor (unsatisfactory) result, according to the Mayo elbow performance index (see appendix).
Woundhealing | 12 months
  Clinical reassessment at Routine follow-ups at every study visit
  - Classification in normal or delayed/impaired. Signs for im-pairment are local secretion, swelling, reddening or wound dehiscence.
Clinical fracture consolidation after one year | 12 months
  Clinical reassessment at Routine follow-ups at every study visit
  - Clinical signs for good consolidation are: no pain while palpating the fracture site.

CONTACTS AND LOCATIONS:
Locations (1):
- Childres Hospital of Eastern Switzerland, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No